CLINICAL TRIAL: NCT05274646
Title: Impact on Risk Stratification of Overlap Syndrome Phenotype (Brugada and Long QT Type 3) in Patients With E1784K Mutation in SCN5A
Brief Title: Impact on Risk Stratification of Overlap Syndrome Phenotype in Patients With E1784K Mutation in SCN5A
Acronym: RISKOVER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/36
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Long QT Syndrome; Brugada Syndrome; Cardiac Conduction System Disease; Arrhythmias, Cardiac
Keywords: Long QT syndrome type 3; Brugada Syndrome; SCN5A gene; E1784K mutation; Cardiac arrhythmias; Cardiac conduction system disease; phenotypic overlap; overlap syndrome; sodium channelopathie
MeSH Terms: conditions — Long QT Syndrome; Brugada Syndrome; Cardiac Conduction System Disease; Arrhythmias, Cardiac; Long QT syndrome type 3; Long Qt Syndrome 3

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- E1784K (glu1784lys) in SCN5A expressing either Long QT syndrome type 3 or Brugada syndrome
- E1784K (glu1784lys) in SCN5A expressing both syndromes (Long QT syndrome and Brugada syndrome)

SUMMARY:
In patients expressing the SCN5A-E1784K mutation (Glu1784Lys), cardiovascular risk is difficult to define as the stratification of these patients is challenging. From our experience, major cardiovascular events (MCE) tend to occur more frequently in patients expressing overlap syndrome phenotype (Brugada syndrome and Long QT syndrome type 3)than in patients expressing a single phenotype (whether Brugada syndrome or Long QT syndrome type 3). This trials is led on the impact on Risk Stratification of Overlap Syndrome Phenotype in Patients With E1784K Mutation in SCN5A ( RISKOVER )

DETAILED DESCRIPTION:
Study design: This study will compare the occurrence of MCE between patients with overlap syndrome phenotype and patients with a single phenotype (whether Brugada syndrome or Long QT syndrome type 3) in a cohort of patients 12 years of age and older with the SCN5A-E1784K mutation. Eligible patients will be identified nationwide and included retrospectively and prospectively. Occurrence of MCE between the group " overlap syndrome " and the group " single phenotype " will be compared.

ELIGIBILITY:
Inclusion Criteria:

* genotype E1784K (glu1784lys) in SCN5A gene

Exclusion Criteria:

* none

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with hereditary cardiac disease
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of MCE | at inclusion
  occurrence of syncop, sudden cardiac death, ventricular arrhythmia, cardiopulmonary arrest collected by a series of medical questions

CONTACTS AND LOCATIONS:
Overall Officials: Maxime CHURET, MD, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de La Réunion, Saint-Pierre, France, Reunion

IPD SHARING:
Plan to Share IPD: No